CLINICAL TRIAL: NCT05796557
Title: ECMO Hemostatic Transfusions in Children
Acronym: ECSTATIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Weill Medical College of Cornell University (Other); University of Utah (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Columbia University (Other); Virginia Commonwealth University (Other); University of Rochester (Other); Children's Hospital and Health System Foundation, Wisconsin (Other); Duke University (Other); Johns Hopkins All Children's Hospital (Other); University of Iowa (Other); Emory University (Other); Schneider Medical Children's Center, Israel (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000034604; 1R34HL159119-01A1 (NIH)
Record Dates: First submitted 2023-03-17; First posted 2023-04-03 (Actual); Results first posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Extracorporeal Membrane Oxygenation Complication; Hemorrhage; Thromboembolism; Transfusion Adverse Reaction
Keywords: Platelet transfusion; ECMO; Bleeding; Clotting; Mortality
MeSH Terms: conditions — Hemorrhage; Thromboembolism; Thrombosis | interventions — Platelet Transfusion

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1 ratio to either arm. Subjects will be stratified by type of extracorporeal membrane oxygenation (ECMO) support (Veno-Arterial vs Veno-Venous), by site, and by age (≤28 days vs >28 days).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and Outcome Assessors will be masked to the intervention, but the clinical team at the bedside will need to know the allocation to be able to prescribe platelet transfusion according to the randomized threshold.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Higher platelet transfusion strategy (Active Comparator): Participants randomized to this arm will be transfused if the platelet count is < 90 x 10e9 cells/L.
  Interventions: Biological: Platelet Transfusion
- Lower platelet transfusion strategy (Experimental): Participants randomized to this arm will be transfused if the platelet count is < 50 x 10e9 cells/L.
  Interventions: Biological: Platelet Transfusion

INTERVENTIONS:
Biological: Platelet Transfusion — Participants will be transfused according to the assigned threshold for each group, with a transfusion dose of 10 mL/kg, up to one adult unit.

SUMMARY:
Critically ill children supported by extracorporeal membrane oxygenation (ECMO) receive large volumes of prophylactic platelet transfusions to prevent bleeding. However, mounting evidence has demonstrated significant morbidity and mortality associated with these transfusions. The ECmo hemoSTAtic Transfusions In Children (ECSTATIC) pilot trial will test two different platelet transfusion strategies, based on two different platelet counts thresholds, one high (higher platelet transfusion strategy) and one low (lower platelet transfusion strategy). The pilot will gather the necessary information to perform a full trial which will provide a better understanding of how to transfuse platelets to children supported by ECMO and reduce the associated morbidity.

DETAILED DESCRIPTION:
Due to coagulopathy and thrombocytopenia induced by hemodilution and the extracorporeal circuit itself, children supported by extracorporeal membrane oxygenation (ECMO) are at significant risk of bleeding. In order to prevent bleeding, pediatric intensivists often prescribe prophylactic platelet transfusions. However, in observational studies, prophylactic platelet transfusions to children on ECMO have been independently associated with increased thrombosis, mortality, and paradoxically, increased bleeding. Guidelines to direct platelet transfusions in this patient population are limited by the lack of evidence and therefore based on expert opinion alone. Given the significant associated risks, it is crucial to provide evidence to guide clinicians.

The ECSTATIC pilot, a randomized controlled trial endorsed by BloodNet, PediECMO, the Extracorporeal Life Support Organization (ELSO), and the Pediatric Acute Lung Injury and Sepsis Investigators (PALISI), will be conducted in ten sites (9 in the US and 1 in Israel). The investigators will enroll an anticipated 50 consecutive critically ill children (0 to <18 years of age), admitted to a participating pediatric, neonatal, or cardiac intensive care unit (PICU/NICU/CICU), on ECMO, and who have either no bleeding or minimal bleeding.

Non-bleeding children 0 to less than 18 years of age will be randomized 1:1 to either a platelet transfusion threshold of 90 x10e9/L (higher platelet transfusion strategy) or 50 x10e9/L (lower platelet transfusion strategy). Participants will be followed until progression to severe bleeding and/or severe thrombosis, decannulation from ECMO, or reach 21 days.

In this pilot, the investigators will test the separation between the lower and higher transfusion strategies. The primary outcomes will be the separation between pre-transfusion platelet counts, and the total platelet dose (in mL/kg/run). Secondary outcomes will be feasibility of patient enrollment and ability for an adjudication committee to determine the severity of bleeding and thrombotic outcomes.

The purpose of this pilot study is to determine the feasibility of the transfusion strategies, intervention parameters, subject availability, and other information regarding outcomes that are essential to complete the design of a large randomized controlled trial.

The large future trial will evaluate the efficacy of the two transfusion strategies, in terms of progression to severe bleeding and/or severe thrombosis. To adequately calculate the sample size, the investigators need to know the difference between the pre-transfusion platelet counts, the screening and inclusion rates, the proportion of patients who are consented within the first 24 hours after cannulation, the proportion of transfusions that are compliant with each arm's strategy, and the number of temporary suspensions.

The proposed pilot trial is innovative in that it is focused on children supported by ECMO, a population in whom transfusion strategies have never been tested previously; it involves the largest separation between the two arms of any platelet transfusion trial conducted in the past; and it involves two newly developed definitions of bleeding and thrombosis particularly applicable to children supported by ECMO.

The pilot trial will provide necessary and sufficient information to proceed with the definitive ECSTATIC Randomized Controlled Trial (RCT) to evaluate the impact of a lower prophylactic platelet transfusion threshold on the clinical outcomes in children on ECMO. ECSTATIC has the potential to optimize efficacy, to reduce platelet transfusion exposure and to decrease mortality and morbidity of these extremely ill infants and children.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill children (0 to <18 years of age)
* Admitted to a participating pediatric, neonatal, or cardiac intensive care unite (PICU/NICU/CICU)
* On extracorporeal Membrane Oxygenation (ECMO)
* Who have either no bleeding or minimal bleeding, within 24 hours of cannulation. Minimal bleeding is defined as:

  * streaks of blood in endotracheal tube or during suctioning only
  * streaks of blood in nasogastric tube
  * macroscopic hematuria
  * subcutaneous bleeding (including hematoma and petechiae) < 5 cm in diameter
  * quantifiable bleeding < 1mL/kg/hr (e.g., chest tube)
  * bloody dressings required to be changed no more often than each 6hr, or weighing no more than 1mL/kg/hr if weighed, due to slow saturation

Exclusion Criteria:

* Post-conception age < 37 weeks at time of screening
* Underlying oncologic diagnosis (defined as receipt of chemotherapy or radiation in the last six months) or recipient of bone marrow transplant in the last year
* Congenital bleeding disorder
* Pregnant or admitted post-partum
* Decision to withdraw or withhold some critical care or interventions
* Known objection to blood transfusions
* On ECMO for > 24 hours at time of enrollment

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Karam, MD, PhD, Principal Investigator — Yale University; Marianne Nellis, MD, MS, Principal Investigator — NewYork-Presbyterian / Weill Cornell
Locations (10):
- United States (9):
  - Children's Healthcare of Atlanta - Emory, Atlanta, Georgia
  - University of Iowa Health Care, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Morgan Stanley Children's Hospital of New York Presbyterian, New York, New York
  - Komansky Children's Hospital of New York Presbyterian, New York, New York
  - Golisano Children's Hospital, Rochester, New York
  - Duke University School of Medicine, Durham, North Carolina
  - Children's Hospital of Richmond at VCU, Richmond, Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Schneider Children's Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Yes
The proposed research will include data from 50 critically ill subjects who are on extracorporeal life support (ECMO) enrolled at ten participating sites. The final dataset will include demographic and medical information, as well as laboratory data.
  After the investigators' proposed research is complete, each participating site will destroy the key linking this data to protected health information (PHI). Thus, the data will then be completely de-identified. However, the investigators believe that there remains the possibility of deductive disclosure of subjects with unusual characteristics, considering the variety of rare conditions leading to ECMO.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The investigators reserve the right to embargo the data for as long as two years after completion of the project (i.e. fall 2027) in order to allow the investigators' research team to publish additional observations from the data.
Access Criteria: The investigators will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying the data after analyses are completed.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Higher Platelet Transfusion Strategy | Lower Platelet Transfusion Strategy
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Higher Platelet Transfusion Strategy | Lower Platelet Transfusion Strategy | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 0.1 [0 to 0.8] | 0.2 [0 to 3.2] | 0.2 [0.0 to 1.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 12 | 10 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 9 | 18 | 27
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 8 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 11
  Not Hispanic or Latino | 15 | 20 | 35
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 24 | 47
  Israel | 2 | 1 | 3
Cannulation Type [Count of Participants; unit: Participants]
  Veno-venous | 5 | 1 | 6
  Veno-arterial | 20 | 24 | 44

OUTCOME MEASURES:

1. Primary Outcome: Total Platelet Transfusion Dose
Description: The total dose (in mL/kg/day) will be computed by the research team, by dividing the total platelet transfusion volume by the patient's weight at admission and the number of days of intervention.
Time Frame: up to day 21
Measure: Median (Inter-Quartile Range); unit: mL/kg/day
Arm/Group | Higher Platelet Transfusion Strategy | Lower Platelet Transfusion Strategy
Number analyzed (Participants) | 25 | 25
mL/kg/day | 7.4 [0 to 16.6] | 0 [0 to 8.4]

2. Secondary Outcome: Feasibility Assessed by the Screening Rate
Description: Feasibility will be assessed by the number of eligible participants that were screened.
Time Frame: At screening
Population: Number of eligible patients among the patients that were screened.
Measure: Count of Participants; unit: Participants
Groups:
- All Screened Patients: Number of patients that were screened.
Arm/Group | All Screened Patients
Number analyzed (Participants) | 159
Participants | 123

3. Secondary Outcome: Feasibility Assessed by the Inclusion Rate
Description: Feasibility will be assessed by the number of eligible participants that were enrolled.
Time Frame: At screening
Population: Number of eligible patients who were enrolled.
Measure: Number; unit: participants
Groups:
- Number of Eligible Patients: Number of eligible patients (all inclusion criteria, no exclusion criteria)
Arm/Group | Number of Eligible Patients
Number analyzed (Participants) | 123
participants | 50

4. Secondary Outcome: Feasibility Assessed by the Number of Informed Consents Signed in the First 24 Hours Post Cannulation.
Description: Feasibility will be assessed by the number of participants that sign consent within the first 24 hours after ECMO cannulation.
Time Frame: At screening
Population: Number of approached patients who consented.
Measure: Number; unit: participants
Groups:
- Approached Patients: Number of approached patients
Arm/Group | Approached Patients
Number analyzed (Participants) | 80
participants | 50

5. Secondary Outcome: Compliance With Transfusion Thresholds
Description: The proportion of transfusions that were given for platelet counts below the arm threshold will be computed to assess compliance.
Time Frame: up to Day 21
Population: Number of transfusion decisions (either to transfuse or not to transfuse, based on platelet count).
Measure: Number; unit: Compliant transfusion
Units Other Than Participants: Transfusion
Arm/Group | Higher Platelet Transfusion Strategy | Lower Platelet Transfusion Strategy
Number analyzed (Participants) | 25 | 25
Number analyzed (Transfusion) | 319 | 389
Compliant transfusion | 316 | 386

6. Secondary Outcome: Participants With at Least One Temporary Suspension
Description: The number of participants who required at least one temporary suspension during ECMO.
Time Frame: up to Day 21
Measure: Count of Participants; unit: Participants
Arm/Group | Higher Platelet Transfusion Strategy | Lower Platelet Transfusion Strategy
Number analyzed (Participants) | 25 | 25
Participants | 6 | 8

7. Secondary Outcome: Duration for Temporary Suspensions
Description: The investigators will collect information on the duration of each suspension.
Time Frame: up to Day 21
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Higher Platelet Transfusion Strategy | Lower Platelet Transfusion Strategy
Number analyzed (Participants) | 25 | 25
Hours | 7.5 [1.5 to 19.6] | 13.5 [1.8 to 23.7]

8. Secondary Outcome: Progression to Composite Outcome of Severe Bleeding and/or Severe Thrombotic Event
Description: The investigators will collect the proportion of participants who progress to a composite outcome of severe bleeding and/or severe thrombosis. The outcome will be adjudicated by an external review committee, blinded to the allocation arm.
Time Frame: up to Day 21
Measure: Count of Participants; unit: Participants
Arm/Group | Higher Platelet Transfusion Strategy | Lower Platelet Transfusion Strategy
Number analyzed (Participants) | 25 | 25
Participants | 4 | 5

9. Secondary Outcome: Number of Participants Who Were Withdrawn and/or Lost to Follow-up
Description: Number of patients who withdraw from the study and/or are lost to follow-up (i.e., withdraw and/or are missing 90-day mortality assessment)
Time Frame: Up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Higher Platelet Transfusion Strategy | Lower Platelet Transfusion Strategy
Number analyzed (Participants) | 25 | 25
Participants | 2 | 2

10. Primary Outcome: Pre-transfusion Platelet Count
Description: Pre-transfusion platelet count, during intervention
Time Frame: During intervention
Measure: Median (Inter-Quartile Range); unit: 10^9 cells/L
Arm/Group | Higher Platelet Transfusion Strategy | Lower Platelet Transfusion Strategy
Number analyzed (Participants) | 25 | 25
10^9 cells/L | 79 [70 to 86] | 43 [39 to 47]

ADVERSE EVENTS:
Time Frame: From randomization up to 24 hours after the end of the intervention, up to 90 days
Description: Serious adverse events, as evaluated by medical monitor.
Arm/Group | Higher Platelet Transfusion Strategy | Lower Platelet Transfusion Strategy
All-Cause Mortality (participants affected / at risk) | 1/25 | 2/25
Serious Adverse Events (participants affected / at risk) | 4/25 | 5/25
Other Adverse Events (participants affected / at risk) | 5/25 | 5/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Higher Platelet Transfusion Strategy (N=25) | Lower Platelet Transfusion Strategy (N=25)
Bleeding (Blood and lymphatic system disorders) | 3 | 4
Clotting (Blood and lymphatic system disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Higher Platelet Transfusion Strategy (N=25) | Lower Platelet Transfusion Strategy (N=25)
Bleeding (Blood and lymphatic system disorders) | 3 | 4
Clotting (Blood and lymphatic system disorders) | 2 | 0
Accidental Removal of Vascular Access (Surgical and medical procedures) | 0 | 1 — Accidental removal of arterial line, requiring replacement.

LIMITATIONS AND CAVEATS:
No limitations or caveats to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT05796557/Prot_SAP_000.pdf